CLINICAL TRIAL: NCT01401998
Title: Core A: The Hepato/Renal Fibrocystic Diseases Translational Resource (ARPKD Database Study)
Brief Title: ARPKD Database Study
Acronym: ARPKD
Status: Recruiting | Type: Observational
Sponsor: Children's Hospital of Philadelphia (Other)
Collaborators: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Sponsor
Other Study IDs: 19-016284; 2P30DK074038-06 (NIH); NCT00575705 (obsolete NCT alias)
Record Dates: First submitted 2011-07-22; First posted 2011-07-26 (Estimated); Last update posted 2025-06-13 (Actual); Status verified 2025-06

CONDITIONS: Hepato/Renal Fibrocystic Disease; Autosomal Recessive Polycystic Kidney Disease; Joubert Syndrome; Bardet Biedl Syndrome; Meckel-Gruber Syndrome; Congenital Hepatic Fibrosis; Caroli Syndrome; Oro-Facial-Digital Syndrome Type I; Nephronophthisis; Glomerulocystic Kidney Disease
Keywords: cystic kidney disease; polycystic kidney disease; congenital hepatic fibrosis; genetic disease
MeSH Terms: conditions — Polycystic Kidney, Autosomal Recessive; Agenesis of Cerebellar Vermis; Bardet-Biedl Syndrome; Meckel syndrome type 1; Hepatic Fibrosis, Congenital; Caroli Disease; Nephronophthisis, familial juvenile; Kidney Diseases, Cystic; Polycystic Kidney Diseases; Genetic Diseases, Inborn

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Biospecimen Retention: Samples With DNA — Blood-derived DNA and lymphocytes for EBV-immortalized cell lines. Remnant tissue samples affected with Hepato/Renal Fibrocystic Diseases
Oversight: Data Monitoring Committee: Yes

SUMMARY:
Hepato-renal fibrocystic diseases (HRFD) is a term developed that encompasses rare diseases such as Autosomal Recessive Polycystic Kidney Disease (ARPKD), and other diseases with common features (Joubert syndrome, Bardet Biedl syndrome, Meckel-Gruber syndrome, congenital hepatic fibrosis (CHF), Caroli syndrome (CS), polycystic liver disease, oro-facial-digital syndrome, nephronophithisis (NPHP), and glomerulocystic Kidney Disease).

The lack of enough routinely available resources for these diseases to be well diagnosed and treated, would be best resolved by coordinated case accrual and sharing of clinical data and bio-specimens (DNA and tissues) among participating institutions, thereby leading to the centralization and sharing of clinical and genetic information, as well as bio-materials, providing an important engine for more rapid research progress and community understanding through the creation of research networks.

This study aims to build a registry of a clinical database (medical health information), a mutational database (genetic information) and an educational resource about HRFD to eventually provide information about these diseases to families, physicians and genetic counselors via our existing HIPAA- approved study website.

Goals for the Core A: The Hepato/Renal Fibrocystic Diseases Translational Resource are:

1. - Clinical Database:

   • Expand our comprehensive Clinical Database to include information from all patients who meet the inclusion criteria for hepato/renal fibrocystic diseases.
2. - Mutational Database:

   * Test children with ARPKD and other hepato/renal fibrocystic disease to identify genetic mutations, establish a DNA bank for patients with hepato/renal fibrocystic diseases and develop a Mutational Database. This Database will be capable of linking clinical and mutational information via a unique identifier in a searchable format to facilitate genetic research (e.g. genotype-phenotype correlations, new disease gene studies, and modifier gene studies), translational studies, and clinical trials.

     3- Tissue Resource:
   * Much of the research that is performed on diseases of the kidney, including recessive genetic diseases, requires human tissue from both affected as well as non-affected (controls) individuals. In this Core Resource, we are establishing an independent tissue resource which would supply investigators throughout North America with samples of hepato/renal fibrocystic disease affected tissues for studies of these disorders.

     4- Educational Resource:
   * Expand our multi-media, web-based resource to provide a reliable up-to-date, and comprehensive informational resource for ARPKD and Hepato/Renal Diseases families, their physicians, and genetic counselors.

DETAILED DESCRIPTION:
Subject's will have the option of the database, genetic, tissue, and urine section of the study.

This study does not require a clinic visit to our center. We will review past, current, and future medical information related to the database participants. Information that we will collect include: clinic notes, lab results, and physician consult reports. Subjects may be asked to sign a release of medical information form to allow the study team access to their medical records. When the information is received, the research study team will enter medical data into the Hepato-Renal Fibrocystic Diseases (HRFD) clinical database. There will be initial data entry and then annual follow up data entries lasting for the duration of this study or until subjects choose to not participate in the study anymore. We will remove subject's name or any other identifiable health information (such as name, address) from received records before entering medical data into the HRFD clinical database.

If subjects choose to participate in the optional genetic material testing portion of the study, either the referring site may draw the blood sample (~5 mL or a teaspoon) or the research team will send a mailer and a blood collection kit. Samples will be collect from the subject, subject's father, and subject's mother. Once the blood samples are collected, the samples will be sent to Children's Hospital of Philadelphia and each sample will be processed to obtain the DNA. These DNA samples will be labeled only with an identifier that is unique to the subject and stored in the BioRepository at CHOP.

If blood samples are unobtainable from the subject's parents, saliva samples can be collected as an alternative.

In the event of research tissue donation, we will collect tissue (kidney, liver, pancreas, lung, brain, heart, and/or placenta) samples for storage at CHOP Tissue Repository. This tissue repository will be an important source for researchers to access tissue for analysis. Dr. Lisa Guay-Woodford and team will be facilitating the consenting process for collection and storage of tissue as part of her role. For individuals that will be undergoing an autopsy or nephrectomy/hepatectomy, consent will be obtained from the study participants and/or their parents. The Pathology Department at the institution performing the procedures (autopsy or nephrectomy/hepatectomy) will collect tissue according to specified protocol provided by the study coordinator. Upon receipt, the CHOP Repository will process and store the specimens.

Children's Hospital of Philadelphia will serve as a research site to store and process blood specimens, and analyze electronic medical records data via REDcap.

ELIGIBILITY:
Inclusion Criteria:

* Demonstration of hepato/renal fibrocystic disease by clinical information, imaging studies, biopsy, autopsy, or genetic testing.

Exclusion Criteria:

* ADPKD Urinary tract malformations Major congenital anomalies of other systems

Max Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: In view of the genetics and demographics of the recessive disorders comprising the spectrum of hepato/renal fibrocystic diseases, we estimate that 50% of the subjects will be female; that 90% of the subjects will be Caucasian and the remainder will belong to the following racial/ethnic categories: 5% African-Americans; 3% Hispanics; 1% Asians; and 1% or less will be other categories.
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2011-06; Primary Completion 2030-09 (Estimated); Study Completion 2030-12 (Estimated)

PRIMARY OUTCOMES:
Core A: The Hepato/Renal Fibrocystic Diseases Translational Resource (Hepato/Renal Fibrocystic Diseases Core Center (UAB HRFDCC)) | five years
  Core A: The Hepato/Renal Fibrocystic Diseases Translational Resource:
  The aims of this Core are:
  * Expand our current clinical and mutational database and establish a DNA bank
  * Establish a national tissue repository for hepato/renal fibrocystic diseases
  * Broaden the portfolio of educational tools developed for physicians and patients to encompass the hepato/renal fibrocystic diseases spectrum of disorders.
  A unique aspect of this Core is that it builds on established clinical, genotyping, and educational programs and through the P30 mechanism will make these data/resources available to the broader community of interested investigators

CONTACTS AND LOCATIONS:
Overall Officials: Lisa Guay-Woodford, MD, Principal Investigator — Children's Hospital of Philadelphia
Locations (6):
- United States (6):
  - Children's National Hospital, Washington D.C., District of Columbia
  - Emory, Atlanta, Georgia
  - Boston Children's, Boston, Massachusetts
  - Cincinnati Children's, Cincinnati, Ohio
  - Children's Hospital of Philadelphia, Philadelphia, Pennsylvania
  - University of Utah, Salt Lake City, Utah

REFERENCES:
- See also: Core A: The Hepato/Renal Fibrocystic Diseases Translational Resource — https://arpkdb.org/